CLINICAL TRIAL: NCT01451918
Title: Regulation of Intestinal (and Hepatic) Lipoprotein Secretion by Resveratrol
Brief Title: Regulation of Intestinal and Hepatic Lipoprotein Secretion by Resveratrol
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: RESV10-0537-A
Record Dates: First submitted 2011-10-11; First posted 2011-10-14 (Estimated); Last update posted 2014-05-06 (Estimated); Status verified 2012-05

CONDITIONS: Dyslipidaemia; Insulin Resistance
Keywords: Dyslipidaemia; Insulin resistance; Type 2 Diabetes
MeSH Terms: conditions — Dyslipidemias; Insulin Resistance; Diabetes Mellitus, Type 2 | interventions — Resveratrol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Resveratrol (Active Comparator)
  Interventions: Drug: Resveratrol
- Placebo (Placebo Comparator)
  Interventions: Drug: Resveratrol

INTERVENTIONS:
Drug: Resveratrol — 500mg bid for one week followed by 1 gram bid for one week prior to lipoprotein study.

SUMMARY:
Resveratrol, an ingredient of red wine and available in Canada in highly purified form as an over-the-counter health supplement, has been shown to have a number of health benefits. Data from in vitro and animal studies suggest that it has beneficial effects on insulin sensitivity and lipid lowering. The investigators are not aware, however, of any mechanistic studies that have examined the effect of highly purified resveratrol in vivo on lipoprotein metabolism in humans. Given the potential therapeutic benefit of resveratrol in correcting the metabolic abnormalities of insulin resistant individuals the investigators plan to examine the effects of resveratrol on intestinal and hepatic lipoprotein production in humans.

DETAILED DESCRIPTION:
Subjects will receive resveratrol (Transmax 1 x 500mg tablets bid for one week followed by 2 x 500mg bid for the second week (Biotivia Longevity Biologicals, New York, NY, USA) or placebo and advised to start taking the tablets 14 days prior to the first lipoprotein kinetics study.

For the lipoprotein kinetics study subjects will receive an infusion of stable isotope enriched leucine and a bolus of stable isotope enriched glycerol in order to measure the rates of fatty acid synthesis, apolipoprotein and triglyceride turnover respectively. This in vivo stable isotope enrichment methodology has been widely established and used by investigators around the world for more than 30 years to examine the metabolism of various metabolites in humans.

On the first day of the 2 day admission to hospital for the lipoprotein kinetics study, following an overnight fast, at approximately noon on day 1 of the study the subject will be admitted to hospital and will have a 30ml fasting blood sample drawn for analysis of plasma glucose, total plasma cholesterol, LDL-cholesterol, HDL cholesterol, triglycerides (TG), free fatty acids (FFA), insulin, cytokines, stable isotope enrichment and a more detailed analysis of triglyceride rich lipoprotein (TRL) composition (lipid and apolipoprotein content). The subject will be allowed to eat regular meals during the day but will fast overnight after 7pm.

At 4am the subject will begin to ingest the first of 17 identical small hourly aliquots of a liquid formula called Great Shake Plus (Hormel), each hourly dose equivalent to 1/17th of their estimated daily caloric requirement calculated by the Harris-Benedict formula. Apart from the shake the subject will not eat until the end of the study at 7pm that night. This will provide a steady state fed state for the subsequent assessment of lipoprotein turnover kinetics. At 7am 2 iv's will be inserted into a superficial vein in each forearm, one for infusion and one for sampling.

At 7 am (the investigators will refer to this time point as 0hr of the lipoprotein turnover study), the lipoprotein turnover study will begin. An iv bolus of deuterated-glycerol (d5-glycerol, 75 micromol/kg) will be administered, followed by a primed-constant infusion of deuterated leucine (L-[5,5,5-2H3]-leucine; d3-leucine, 98%, Cambridge Isotope Laboratories, Andover, MA, USA)(10 micromol/kg bolus followed by 10 micromol/kg/hr for 10 hours). Blood samples will be collected prior to and at regular time intervals for 10 hours after the iv bolus of d3-glycerol (for 13C-triglyceride palmitate enrichment to assess de novo lipogenesis) and start of the constant infusion of d3-leucine (for assessment of lipoprotein kinetics). Insulin sensitivity will be assessed by calculation of HOMA-IR.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women, aged 23 to 60 years
2. Fasting plasma triglycerides between 2.0 and 5.0 mmol/l
3. Body mass index 25 kg/m2 to 35 kg/m2
4. Minimum body weight 64kg
5. Hemoglobin above 130g/L.
6. Research volunteers must be able to provide informed consent and be willing to comply with protocol requirements.
7. HOMA-IR (a measure of insulin resistance calculated from fasting blood glucose and insulin) >4.0.

   .

Exclusion Criteria:

1. Subject has a history of hepatitis/hepatic disease that has been active within the previous two years.
2. Any significant active (over the past 12 months) disease of the gastrointestinal, pulmonary, neurological, renal (Cr > 1.5 mg/dL), genitourinary, hematological systems, or has severe uncontrolled treated or untreated hypertension (sitting diastolic BP > 90 or systolic >140) or proliferative retinopathy
3. Any dehydration or excessive vomiting
4. History of diabetes or 75g OGTT indicative of diabetes.
5. Cancer or history of cancer
6. Any history of a MI or clinically significant, active, cardiovascular history including a history of arrhythmia's or conduction delays on ECG, unstable angina, or decompensated heart failure.
7. Any active medical illness
8. Any laboratory values: AST > 2x ULN; ALT > 2x ULN TSH>5mU/l or <0.01 mU/l
9. Any clinically relevant abnormal blood/urine screening test results that are outside of the normal reference range and are significant to the investigator will be excluded
10. Any current hormonal disorder or history or hormonal disorders
11. Any bleeding disorders or autoimmune conditions
12. Any allergies to any of the ingredients in the study product or placebo ie: hypersensitivity to resveratrol, grapes, red wine, red wine polyphenols and microcrystalline microcellulose
13. Current addiction to alcohol or substances of abuse as determined by the investigator.
14. Mental incapacity, unwillingness or language barrier precluding adequate understanding or cooperation
15. Taking any prescription or non-prescription medications at the time of the study
16. Taking any natural health products during the course of the study
17. Having donated blood three months prior to and three months post study procedures
18. A pregnancy test will be performed 1 to 3 days prior to each study in all female subjects (visit #4, and visit #7 before taking study drug). Those who test positive for pregnancy will be excluded.
19. If you are breast-feeding or lactating you will be excluded from the study.
20. Women taking the oral contraceptive pill will be excluded from the study.
21. All current smokers or those who have smoked more than 1 pack per day for 5 years or more.
22. Those with ferritin levels below 50 ug/L will be excluded
23. Study Participants who experience serious adverse event or who no longer satisfy the inclusion /exclusion criteria during the trial will be withdrawn

Ages: 23 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2011-10; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Examine the effect of resveratrol on ApoB 100 and ApoB 48 production in humans | 2 weeks
  10 hour lipoprotein turnover study as described above following 2 weeks treatment with resveratrol or placebo.

SECONDARY OUTCOMES:
Assess the change in insulin sensitivity with resveratrol treatment | 2 weeks
  HOMA-IR calculated from fasting insulin and fasting glucose will be used to assess change in insulin sensitivity before and after 2 weeks of resveratrol treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Gary Lewis, MD, Principal Investigator — UHN Toronto
Locations (1):
- Toronto General Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Dash S, Xiao C, Morgantini C, Szeto L, Lewis GF. High-dose resveratrol treatment for 2 weeks inhibits intestinal and hepatic lipoprotein production in overweight/obese men. Arterioscler Thromb Vasc Biol. 2013 Dec;33(12):2895-901. doi: 10.1161/ATVBAHA.113.302342. Epub 2013 Sep 26. PMID 24072699